CLINICAL TRIAL: NCT01638637
Title: Prospective Collection of Female First-catch Urine, Vaginal Swab, Cervical, and Endocervical Swab Specimens and Male Urethral Swab and First-catch Urine Specimens for Testing With the PANTHER® System
Brief Title: Prospective Collection of Female and Male Specimens for PANTHER® System Testing
Status: Completed | Type: Observational
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: AGCPS-US11-002; AC2PS-US12-001 (Other: Gen-ProbeAC2PS-US12-001Eval of COMBO2 Assay On PANTHER System in Male Urine is testing protocol for AGCPS-US11-002)
Record Dates: First submitted 2012-02-29; First posted 2012-07-12 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Chlamydia Infections; Gonorrhea
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Specimen Collection
  Interventions: Device: APTIMA Assays; PANTHER System

INTERVENTIONS:
Device: APTIMA Assays; PANTHER System — APTIMA Assays; PANTHER System
  Other Names: APTIMA Combo, APTIMA CT, APTIMA GC

SUMMARY:
The objective of this study is to obtain female first-catch urine, vaginal, cervical and endocervical swabs and male first-catch urine and urethral swabs for testing with multiple APTIMA Assays on the Gen-Probe PANTHER® System

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 16 years of age at the time of enrollment and is currently sexually active (has had intercourse within the past 12 months)
* The subject and/or legally authorized representative is willing to undergo the informed consent process prior to study participation (a minor will need the documented consent of his/her parent or legal guardian, unless the site has an institutional review board (IRB)-approved waiver for parental consent for minors)

In addition, the subject must meet at least one of the following criteria:

* The subject reports symptoms consistent with a suspected STI such as abnormal discharge, genital itching, pain/discomfort during sexual intercourse or urination, and/or lower abdominal discomfort
* Subject is asymptomatic and known to be partners with, or a contact of, a person with a confirmed or suspected STI(s)
* Subject is asymptomatic and undergoing screening evaluation for possible STIs
* Subject (female) is asymptomatic and undergoing a routine examination with a pelvic examination

Exclusion Criteria:

* A potential subject will be ineligible for clinical trial enrollment if the subject, clinician, or medical record reports any of the following:
* The subject took antibiotic medications within the last 21 days
* Subject already participated in this study
* Subject has a history of illness that the principal investigator (PI) or designee considers could interfere with or affect the conduct, results, and/or completion of the clinical trial
* Subject has a history of illness that the PI or designee considers could create an unacceptable risk to the subject if enrolled

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Symptomatic and asymptomatic subjects at least 16 years of age.
Sampling Method: Probability Sample
Enrollment: 1492 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Qualitative detection of ribosomal RNA from Chlamydia trachomatis and/or Neisseria gonorrhoeae (GC) to aid in the diagnosis of chlamydial and/or gonococcal urogenital disease | approximately one year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reid, PhD, Study Director — Gen-Probe, Incorporated
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Anthony Mills MD Inc., Los Angeles, California
  - Benchmark Research, San Francisco, California
  - Planned Parenthood Southern New England, New Haven, Connecticut
  - AGA Clinical Trials, Hialeah, Florida
  - Wishard Health Services, Indianapolis, Indiana
  - Louisiana State University Health Sciences, New Orleans, Louisiana
  - John Hopkins University, Baltimore, Maryland
  - New England Center for Clinical Research - New Bedford Clinic, New Bedford, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Laboratory Corporation of America, Burlington, North Carolina
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Molecular Pathology Laboratory Network, Inc., Maryville, Tennessee
  - Planned Parenthood Houston and Southeast Texas, Houston, Texas
  - Tidewater Clinical Research, Inc. -Tidewater Physicians for Women, Norfolk, Virginia